CLINICAL TRIAL: NCT02371798
Title: Diagnosing Endolymphatic Hydrops in Patients With Meniere Disease Using Magnetic Resonance Imaging With Intravenous Gadolinium Administration
Brief Title: Unilateral Meniere Disease: Can Double Dose Gadolinium and Delayed Imaging Make the Diagnosis?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Patricia Hudgins, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00077659
Record Dates: First submitted 2015-02-19; First posted 2015-02-26 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Meniere Disease
MeSH Terms: conditions — Meniere Disease | interventions — Gadolinium DTPA

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Double dose of Gadopentetate dimeglumine (Experimental): Subjects with a clinical diagnosis of unilateral Meniere Disease (MD) will undergo 3T MR imaging with a double dose of intravenous (IV) gadolinium contrast injection: 0.2 mmol/kg of Gd-DTPA (Magnevist)
  Interventions: Drug: Gadopentetate dimeglumine

INTERVENTIONS:
Drug: Gadopentetate dimeglumine — IV administration of 0.2 mmol/kg of Gd-DTPA
  Other Names: Magnevist; Gadopentetic acid

SUMMARY:
The purpose of this research study is to see if magnetic resonance imaging (MRI) with a double dose of contrast, or dye, and delayed imaging with MRI can help to diagnose Meniere Disease.

DETAILED DESCRIPTION:
Meniere's disease (MD) is a medical condition causing attacks of vertigo, ringing in the ears, hearing loss and often a fullness in the ear. Currently there is no definitive test to diagnose the problem. It is believed to be caused by inner ear abnormalities, specifically of an over-collection of lymphatic fluid.The goal of this trial is to determine if an MRI with double dose of IV gadolinium can be diagnostic.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unilateral Meniere Disease (MD) per the Committee on Hearing and Equilibrium of the American Academy of Otolaryngology-Head and Neck Surgery (AAO-HNS)
* Glomerular filtration rate (GFR) > 90 mls/min/1.73 m2
* Creatinine (Cr) level serum < 1.6 mg/dl

Exclusion Criteria:

* Age < 18 years
* Diagnosis of bilateral MD
* History of prior temporal bone surgery
* History of cochlear implant placement
* Pacemaker, cardiac implantable electronic device, shrapnel, aneurysm clips or other metal objects that are prohibited in the MR suite
* GFR < 90 mls/min/1.73m2
* Cr level > 1.6 mg/d
* Lack of IV access
* Contrast allergy to gadolinium agent
* Pregnancy
* Claustrophobia necessitating parenteral anxiolytics
* Patients who are unable to provide informed consent for themselves

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Grade of endolymphatic hydrops (EH) in the cochlea and vestibule | 6 hours after intravenous contrast injection
  Two Certificate of Added Qualifications (CAQ)-certified neuroradiologists will evaluate the MRI findings. The degree of EH in the vestibule and cochlea will be classified as "none", "grade I" and "grade II," with grade I being defined as mild and grade II being defined as significant.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Hudgins, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Department of Otolaryngology Clinic, Atlanta, Georgia, United States